CLINICAL TRIAL: NCT03015207
Title: A Randomised, Double-blinded, Single-dose, Dose-escalation, First Human Dose Trial Investigating Safety, Tolerability and Pharmacokinetics of NNC0194-0499 in Male Subjects With Overweight or Obesity
Brief Title: First Human Dose Trial Investigating Safety, Tolerability and Pharmacokinetics of NNC0194-0499 in Male Subjects With Overweight or Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NN9499-4277; U1111-1181-9045 (Other: WHO)
Record Dates: First submitted 2017-01-06; First posted 2017-01-09 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NNC0194-0499 (Experimental): Injected s.c. /subcutaneously (under the skin)
  Interventions: Drug: NNC0194-0499
- Placebo (Placebo Comparator): Injected s.c. /subcutaneously (under the skin)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NNC0194-0499
  Arms: NNC0194-0499
Drug: Placebo
  Arms: Placebo

SUMMARY:
This trial is conducted in The United States of America. The aim of this trial is to investigate Safety, Tolerability and Pharmacokinetics (the exposure of the trial drug in the body) of NNC0194-0499 in Male Subjects with Overweight or Obesity.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 22-55 years (both inclusive) at the time of signing informed consent
* Body mass index (BMI) between 25.0 and 34.9 kg/m^2 (both inclusive). Overweight should be due to excess adipose tissue, as judged by the investigator

Exclusion Criteria:

* Any concomitant illness or disorder, which in the investigator's opinion might jeopardise the subject's safety or compliance with the protocol
* Subjects aged above or equal to 40 years with an estimated 10-year atherosclerotic cardiovascular disease (ASCVD according to ACC/AHA (American College of Cardiology /American Heart Association) guideline) risk above or equal to 5%
* Male subjects who are not sexually abstinent or surgically sterilised (vasectomy) and are sexually active with female partner(s) and who are not using a highly effective method of contraception (such as condom with spermicide) combined with a highly effective method of contraception for their non-pregnant female partner(s) (Pearl Index below 1%, such as implants, injectables, oral contraceptives, intrauterine devices, diaphragm or cervical cap+spermicide), and/or intend to donate sperm in the period from screening (visit 1) until 3 months following administration of the investigational medical product
* Use of prescription or non-prescription medicinal products including herbal products and non-routine vitamins, within 2 weeks prior to screening, with the exception of occasional use of acetaminophen, ibuprofen or acetylsalicylic acid

Ages: 22 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2017-10-26 (Actual); Study Completion 2017-10-26 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events (TEAEs) | From time of administration of NNC0194-0499 (day 1) to completion of the post-treatment period at follow-up (day 36)

SECONDARY OUTCOMES:
The area under the NNC0194-0499 serum concentration-time curve after a single subcutaneous administration | From pre-dose (day 1) until the followup (day 36)
The maximum concentration of NNC0194-0499 in serum after a single subcutaneous administration | From pre-dose (day 1) until the followup (day 36)
The time to maximum concentration of NNC0194-0499 in serum after a single subcutaneous administration | From pre-dose (day 1) until the followup (day 36)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR,1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, San Antonio, Texas, United States

REFERENCES:
- [Derived] Dahl K, Friedrichsen MH, Ribel-Madsen R, Hansen JS, Clausen JO, Axelsen M, Palle MS, Lippert SL, Bjorkdahl O, Toubro S, Key C, Andersen B. Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of the Novel Long-Acting FGF21 Analog Zalfermin. Clin Transl Sci. 2025 Dec;18(12):e70435. doi: 10.1111/cts.70435. PMID 41351276